CLINICAL TRIAL: NCT06829927
Title: The Effect of E-Booklet Traınıng Created Wıthın the Scope of Comfort Theory on Self-Effıcacy and Comfort Levels in Patıents Wıth Urınary Catheter: a Randomızed Controlled Study
Brief Title: The Effect of E-Booklet Traınıng on Self-Effıcacy and Comfort Level in Patıents Wıth Urınary Catheter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Collaborators: TOGÜ (Unknown)
Responsible Party: Principal Investigator, Şeyda KAZANÇ, Öğr. Gör. Dr., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TOGÜ; Hülya KOÇYİĞİT KAVAK (Other: cUMHURİYETU)
Record Dates: First submitted 2024-07-19; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-09

CONDITIONS: Urinary Catheter
Keywords: urinary cathether; comfort; self-efficiaty

STUDY DESIGN:
Intervention Model Description: This study was planned as a Randomized Controlled Trial to determine urinary catheter-related self-efficacy and comfort levels of patients hospitalized in a university hospital.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind method will be used in the study. Participants will not know which group they are assigned to and statistics will be performed by an independent person to minimize the risk of bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Patients in the control group will not be given any content and their routine care and education will continue. Patients in the control group will be asked to complete the Urinary Catheter Self-Efficacy Scale and Comfort Scale at the 6th and 24 th hours following urinary catheter insertion.
- intervention group (Active Comparator): Patients in the intervention group will be informed about the urinary catheter by the researcher after catheter insertion, and the link to the e-booklet will be given and the patients will be asked to review it. Patients will be asked to fill out the Urinary Catheter Self-Efficacy Scale and Comfort Scale at the 6th and 24th hour following urinary catheter insertion. After the completion of the study, the link to the e-booklet will be given to the patients in the control group to maintain the principle of equality. The research data will be collected by the researcher between 30.09.2024 and 30.10.2025 via Google survey.
  Interventions: Behavioral: e-book

INTERVENTIONS:
Behavioral: e-book — Patients with pilot application will not be included in the study. Patients who agree to participate in the study will be informed by the researcher about the purpose and process of the study, and their written and verbal informed consent will be obtained. Patients will be informed that the decision on whether or not to participate in the study is entirely their own, that no money will be deducted from their health insurance or any money will be paid to them, that the data to be collected from this study will only be used within the scope of the research, and that confidentiality will be strictly ensured. Pretests (Personal Information Form, Urinary Catheter Self-Efficacy Scale and Comfort Scale) will be administered to the patients whose consent is obtained.
  Arms: intervention group

SUMMARY:
Urinary catheterization is the insertion of a tube through the urethra into the bladder to empty or flush the bladder. Catheterization is preferred in patients with urinary retention and urinary incontinence, in patients who will undergo surgical intervention or in cases where a procedure needs to be performed in the urinary tract, and is applied for short (1-7 days), medium (7-28 days) and long term (longer than 28 days) (National Institute of Diabetes and Digestive and Kidney Diseases. (2023). Urinary catheterization is frequently preferred in applications related to treatment and care. According to the CAUTI report, the frequency of urinary catheterization in hospitalized patients in one year is between 15-25% in the world. This rate is between 10-15% in developed countries and 20-30% in developing countries (CAUTI, 2015).

DETAILED DESCRIPTION:
Urinary catheterization is generally preferred for short-term care and treatment (Clarke et al., 2020; Cutinho et al., 2018). Urinary catheterization is critical in routine health care and can cause many complications such as urinary tract infection, epididymitis, catheter obstruction, trauma, pain, bladder spasm, and hematuria if not used appropriately.Darbyshire et al. (2016) found that 32% of patients experienced leakage, 26% experienced pain, 26% experienced discomfort and 24% experienced obstruction.In fact, it is estimated that 450,000 people in the UK undergo short-term urinary catheterization and complications related to urinary catheter use cause 2100 deaths annually (Feneley et al., 2015).

Although urinary tract infection due to catheterization is common, patients' failure to perform appropriate behaviors and practices related to catheterization causes the infection to progress and the treatment process to be prolonged.Urinary tract infections account for approximately 20% of healthcare-acquired infections in acute care facilities and more than 50% in long-term care facilities (Zegeye et al., 2023). In the United States, urinary tract infections account for 32% of all hospital-acquired infections and are the most common type of hospital-acquired infection, with approximately 449,000 cases of urinary tract infections and an estimated cost of $450 million per year (Abiodun, 2018). In cases where they are not inserted under appropriate conditions, care is not provided effectively and treatment protocols are not followed, they pave the way for the development of resistant microorganisms. Accordingly, urinary tract infection, which requires a long treatment process in patients, causes many negative consequences, including prolonged hospital stay, increased in-hospital mortality and increased health care costs (Anderson et al., 2021; Cutinho et al., 2018; Snyder et al., 2023).

ELIGIBILITY:
Inclusion Criteria:

Patients who can actively use information technologies such as phones and tablets

* Inpatients in the Urology Clinic
* Conscious and oriented patients
* Patients aged 18-75 years
* Patients with short-term catheterization
* Patients without hearing and communication disabilities
* Literate patients

Exclusion Criteria:

* Patients who incompletely completed the data collection tool
* Patients with hearing, vision and comprehension problems,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
First Follow-up (Personal Information Form, Urinary Catheter Self-Efficacy Scale and Comfort Scale | after catheterization ( First 1 hour)
  Pretest (Descriptive statistics will be shown with frequencies and percentages, and the distribution of variables according to scale scores will be shown with median (minimum-maximum) values.

SECONDARY OUTCOMES:
Second Follow-up (Urinary Catheter Self-Efficacy Scale and Comfort Scale) | 6 hours
  Second Follow-up . The conformity of the data to normal distribution will be evaluated by Kolmogrov Smirnow test and Mann-Whitney U and Kruskal-Wallis tests, which are non-parametric tests, will be used to compare variables that do not conform to normal distribution. Normally distributed data will be evaluated with t test and Anova test. In order to determine the differences in variables with more than two groups, the Dunn-Bonferroni test from Post-Hoc tests will be used. The relationship between self-efficacy and comfort level will be determined by Spearman Correlation Coefficient. Significance level p<0.05 will be taken in the tests.
Third Follow-up(Urinary Catheter Self-Efficacy Scale and Comfort Scale) | 24 Hours
  Third Follow-up . The conformity of the data to normal distribution will be evaluated by Kolmogrov Smirnow test and Mann-Whitney U and Kruskal-Wallis tests, which are non-parametric tests, will be used to compare variables that do not conform to normal distribution. Normally distributed data will be evaluated with t test and Anova test. In order to determine the differences in variables with more than two groups, the Dunn-Bonferroni test from Post-Hoc tests will be used. The relationship between self-efficacy and comfort level will be determined by Spearman Correlation Coefficient. Significance level p<0.05 will be taken in the tests.

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Koçyiğit KAVAK, Study Chair — Cumhuriyet University; Şerife Karagözoğlu, Prof. Dr., Principal Investigator — Cumhuriyet University
Locations (1):
- Tokat Gaziosmanpaşa University, Tokat/Merkez, Tokat Province, Turkey (Türkiye)